CLINICAL TRIAL: NCT05784181
Title: Bipolar Versus Laser Enaculation of Prostate for >80gram Prostate .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hossam Kandeel, Yassin Abdel Ghaffar St- from Gamal Abdel Anasar St - Faculty of Medicine., Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2-2022
Record Dates: First submitted 2022-02-08; First posted 2023-03-24 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Bipolar TURP , Laser Enucleation in Management of Enlarged Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- patients prostatic volume more than 80 gm turp by bipolar resection (Other): pt with 80gm prostate size underwent bipolar resection
  Interventions: Device: bipolar transurethral resection and Laser enaculation by holmium: YAG laser
- patients prostatic volume more than 80 gm turp by Laser enaculation by holmium: YAG laser (Other): pt with 80gm prostate size underwent Laser enaculation by holmium: YAG laser
  Interventions: Device: bipolar transurethral resection and Laser enaculation by holmium: YAG laser

INTERVENTIONS:
Device: bipolar transurethral resection and Laser enaculation by holmium: YAG laser — Laser enaculation by holmium: YAG laser

SUMMARY:
Transurethral resection of the prostate (TURP ) still the gold standerad for surgical management of enlarged prostate .However , many minimally invasive procedures are now in the comparative track with Bipolar resection as Laser enaculation.

Holmium laser prostatectomy was introduced since 1994 . different types of uses by laser were introduced either resection or enaculation with good outcomes and less complications .

One of the most important issues related to large prostate management is the retreatment after Bipolar resection , another issue that prolonged catheter time post resection .

DETAILED DESCRIPTION:
Transurethral resection of the prostate (TURP ) still the gold standerad for surgical management of enlarged prostate .However , many minimally invasive procedures are now in the comparative track with Bipolar resection as Laser enaculation.

Holmium laser prostatectomy was introduced since 1994 . different types of uses by laser were introduced either resection or enaculation with good outcomes and less complications .

One of the most important issues related to large prostate management is the retreatment after Bipolar resection , another issue that prolonged catheter time post resection , so , we try to analyze the effect of Laser enaculation of the prostate in comparison to Bipolar resection in prostate more than 80 gm .

Aim of the work:

Aim of the work is to compare the efficacy of Bipolar versus Laser enaculation of prostate for >80gram.

Patients and Methods:

A randomized comparative study will be conducted at Menoufia university hospital , urology department. patients will be selected after informed consent.

Inclusion criteria: similar for all patients prostatic volume more than 80 gm , peak urinary ﬂow rate measurement (Qmax) <15 ml/s, International Prostate Symptom Score (IPSS) of >8 , postvoid residual (PVR) <400 ml.

Exclusion criteria: Patients with prostate size less than 80gm , urethral stricture, acute urinary tract infection, repeated treatment .

Preoperatively, all the patients will undergo thorough process of history taking , clinical examination, and investigations in the form of abdominopelvic and trans rectal ultrasonography , PSA ,urine analysis, urine culture if needed and routine pre-operative lab investigations as (CBC , PT, LFTs, serum creatinine and RBS).

The treatment modality chosen for an individual will be randomized . All patients with positive urine culture will be treated by proper antibiotics before the procedures.

Peri-operatively , all patients will receive a single shot of pre-operative antibiotic.

For the first group patients transurethral resection of prostate For the second group patients Laser enaculation by holmium: YAG laser Postoperatively, patients will undergo IPSS score , flowmetry post operative after 3months .

ELIGIBILITY:
Inclusion Criteria:

- similar for all patients prostatic volume more than 80 gm , peak urinary ﬂow rate measurement (Qmax) <15 ml/s, International Prostate Symptom Score (IPSS) of >8 , postvoid residual (PVR) <400 ml

Exclusion Criteria:

* Patients with prostate size less than 80gm , urethral stricture, acute urinary tract infection, repeated treatment .

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
compare the efficacy of Bipolar versus Laser enaculation of prostate for >80gram. | 1 year
  compare the efficacy of Bipolar versus Laser enaculation of prostate for >80gram.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Menoufia -, Egypt